CLINICAL TRIAL: NCT06106347
Title: Analysis of Visual and Ocular Outcomes of Computer Vision Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Refaat Refaee, Resident of ophthalmology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-10-02MS
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CVS group: positive CVS diagnosis
  Interventions: Device: mfERG device (RETIscan; Roland Instruments, Wiesbaden, Germany)
- control: participants with no-CVS diagnosis
  Interventions: Device: mfERG device (RETIscan; Roland Instruments, Wiesbaden, Germany)

INTERVENTIONS:
Device: mfERG device (RETIscan; Roland Instruments, Wiesbaden, Germany) — physiological macular function

SUMMARY:
The digital technology is universal and has spread worldwide; thus, digital behaviour has dramatically changed peoples' lifestyles. Previous studies have reported that individuals interact with digital screens for up to 12 hours daily,1,2 and the American Optometric Association defined a combination of ocular and extraocular symptoms that affects the screen users as computer vision syndrome (CVS).3 However, our current understanding of digital technology and its harmful impact on the eye and public health,1,4,5 visual performance,6-8 sleep patterns,7,8 circadian rhythms,5,8 musculoskeletal system activities,3,4 and underlying physiological mechanisms9 remains incomplete and is associated with misconceptions.1 Therefore, educational programs that include protective measures and health campaigns are necessary.10 Computer vision syndrome (CVS) is also called with other names as digital eye strain (DES),3 occupational asthenopia, digital asthenopia,1 and video display terminal syndrome (VDTS). CVS ocular symptoms include visual blur with an underlying mechanism that is not fully understood,10 dry eye disease (DED),3 eye redness and irritation, eyestrain, fatigue, discomfort, difficulty in refocusing the eyes, and diplopia.3,4. CVS extraocular symptoms include headache, sleep disturbances, depression,7,8 musculoskeletal aches, such as neck/shoulder/back pain, difficulty in writing or holding objects, pain in thumbs, fingers, or wrists because of tendonitis and/or arthritis.

Smartphones are used extensively worldwide by people of all ages, and have close-viewing distance, related high-definition resolution, thousands of time-consuming applications and games in stores, and 24/7 Internet connectivity.

The decline in visual acuity observed in CVS can be attributed to the screen-induced foveal dysfunction11-13 which is a phenomenon that has been extensively documented in the literature using multifocal electroretinogram (mfERG) examinations. Previous studies11-13 consistently reported the presence of this dysfunction, which has been linked to prolonged exposure to digital screens emitting blue light. Notably, recent research has demonstrated noteworthy improvements in foveal responses following a strict reduction in screen time for duration of four weeks.13 These improvements were found to correspond with enhanced visual performances, indicating a positive relationship between the reversal of screen-induced foveal dysfunction and visual outcomes. These findings highlight the reversible nature of screen-induced foveal dysfunction and its potential impact on visual acuity. They support the notion that reducing screen time can serve as an effective intervention strategy, leading to substantial improvements in both foveal responses and overall visual performance.13 The computer vision syndrome questionnaire (CVS-Q) is a self-administered scale that evaluates the frequency and intensity of 16 ocular and visual symptoms related to the use of digital devices. The scoring of the questionnaire follows the procedure of the original version. The 16 items (CVS-symptoms) are scored with two rating scales: one for frequency (never, occasionally, often, or always), and one for intensity (moderate, intense). The responses to the two rating scales for each item are combined multiplicatively into a single scale called symptom severity, and the result should be recoded as 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the worker is considered to suffer computer vision syndrome .14 Ocular surface disease index is a quick self-assessment questionnaire of the symptoms of ocular irritation in dry eye disease (DED) and how they affect functioning related to vision. This 12-item questionnaire assesses dry eye symptoms and the effect it has on vision-related function in the past week of the patient's life.15 The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.15 DED, also known as keratoconjunctivitis sicca, is the condition of having dry eyes. Symptoms include dryness in the eye, irritation, redness, discharge, blurred vision, and easily fatigued eyes. Symptoms range from mild and occasional to severe and continuous. DED can lead to blurred vision, instability of the tear film, increased risk of damage to the ocular surface such as scaring of the cornea, and changes in the eye including the neurosensory system.16

ELIGIBILITY:
Inclusion Criteria:

* include university students and young staff members, 20-30 years old who were spending more than 3 screen-hours daily on average over the last 3 years.

Exclusion Criteria:

* include amblyopia; strabismus; anisometropia; refractive errors higher than 4 D myopia, 4 D hyperopia, or 4 D astigmatism; difference between subjective and cycloplegic refraction >1D; and previous or current systemic or eye disease or surgery.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: include university students and young staff members, 20-30 years old who were spending more than 3 screen-hours daily on average over the last 3 years.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
nV/deg2 | 12 months
  physiological macular function

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

REFERENCES:
- [Background] Vaz FT, Henriques SP, Silva DS, Roque J, Lopes AS, Mota M. Digital Asthenopia: Portuguese Group of Ergophthalmology Survey. Acta Med Port. 2019 Apr 30;32(4):260-265. doi: 10.20344/amp.10942. Epub 2019 Apr 30. PMID 31067419
- [Background] Ahmed SF, McDermott KC, Burge WK, Ahmed IIK, Varma DK, Liao YJ, Crandall AS, Khaderi SKR. Visual function, digital behavior and the vision performance index. Clin Ophthalmol. 2018 Dec 10;12:2553-2561. doi: 10.2147/OPTH.S187131. eCollection 2018. PMID 30573945
- [Background] Iqbal M, Said O, Ibrahim O, Soliman A. Visual Sequelae of Computer Vision Syndrome: A Cross-Sectional Case-Control Study. J Ophthalmol. 2021 Apr 2;2021:6630286. doi: 10.1155/2021/6630286. eCollection 2021. PMID 33868724
- [Background] Iqbal M, Soliman A, Ibrahim O, Gad A. Analysis of the Outcomes of the Screen-Time Reduction in Computer Vision Syndrome: A Cohort Comparative Study. Clin Ophthalmol. 2023 Jan 7;17:123-134. doi: 10.2147/OPTH.S399044. eCollection 2023. PMID 36644605